CLINICAL TRIAL: NCT03545035
Title: Efficacy and Safety in Patients With Chronic Lymphocytic Leukemia (CLL) Treated With Idelalisib and Rituximab in the Clinical Practice: a GIMEMA-ERIC Study
Acronym: LLC178
Status: Completed | Type: Observational
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Collaborators: ERIC Group (Unknown)
Responsible Party: Sponsor
Other Study IDs: LLC1718
Record Dates: First submitted 2018-05-22; First posted 2018-06-04 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; Idelalisib; Rituximab
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — idelalisib; Rituximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: All patients being observed during the study duration.
  Interventions: Drug: idelalisib and rituximab

INTERVENTIONS:
Drug: idelalisib and rituximab — patients with treatment-naïve chronic lymphocytic leukemia (CLL) with TP53 disruption (i.e. 17p- or TP53 mutations) or relapsed/refractory CLL who were treated with idelalisib and rituximab

SUMMARY:
The present study aims at obtaining more in-depth information on how patients with chronic lymphocytic leukemia treated with idelalisib and rituximab react to treatment.

DETAILED DESCRIPTION:
This cohort study will recruit patients with treatment-naïve chronic lymphocytic leukemia (CLL) with TP53 disruption (i.e. 17p- or TP53 mutations) or relapsed/refractory CLL who were treated with idelalisib and rituximab between 01/07/2014 and 31/05/2017 at European centres adhering to the GIMEMA group and the ERIC group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CLL / Small Lymphocytic Lymphoma (CLL/SLL) according to the World Health Organisation (WHO) classification 2008.
* Treatment with idelalisib and rituximab started between the date of Country marketing authorization approval of idelalisib (EMA approval 18/09/2014) and 31/05/2017 given at European centres adhering to the GIMEMA group and the ERIC group.
* One of the two following conditions must be satisfied:

  * Previously untreated CLL requiring therapy according to the NCI criteria (Hallek M et al, Blood 2008)] with deletion 17p13 and/or TP53 mutation.
  * Relapsed refractory CLL., i.e. patients who received at least one previous line of treatment using alkylating agents and/or purine analogues with or without monoclonal antibodies, or high dose steroids requiring therapy according to the NCI criteria (Hallek M et al, Blood 2008)
* Age ≥ 18 years.
* Signed written informed consent, if applicable, according to ICH/EU/GCP and national local law.

Exclusion Criteria:

* Patients with CLL treated with idelalisib within interventional clinical trials or outside the approved indication.
* Patients with:

  * Transformation of CLL to aggressive lymphomas (Richter's Syndrome).
  * HIV infection.
  * Active and uncontrolled HCV and/or HBV infections or liver cirrhosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This cohort study will recruit patients with treatment-naïve chronic lymphocytic leukemia (CLL) with TP53 disruption (i.e. 17p- or TP53 mutations) or relapsed/refractory CLL who were treated with idelalisib and rituximab between 01/07/2014 and 31/05/2017 at European centres adhering to the GIMEMA group and the ERIC group.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2020-10-28 (Actual); Study Completion 2020-10-28 (Actual)

PRIMARY OUTCOMES:
Number of patients responding to treatment | At 12 months from treatment start
  Efficacy profile of idelalisib and rituximab
Number of patients experiencing toxicities | At 12 months from treatment start
  Safety profile of idelalisib and rituximab

SECONDARY OUTCOMES:
Number of patients alive | At 12 months from treatment start
  Overall survival
Number of patients alive without progression of the disease | At 12 months from treatment start
  Progression-free-survival
Number of patients achieving response | At 12 months from treatment start
  Overall response rate

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Cuneo, Study Chair — Ematologia; Azienda Ospedaliera di Ferrara; Gian Matteo Rigolin, Study Director — Ematologia; Azienda Ospedaliera di Ferrara
Locations (38):
- Italy (38):
  - AOU Arcispedale S.Anna - UOC Ematologia e fisiopatologia della coagulazione, Cona, Ferrara
  - Aon Ss. Antonio E Biagio E C. Arrigo - Alessandria - Soc Ematologia, Alessandria
  - Aou Ospedali Riuniti "Umberto I - G.M. Lancisi - G. Salesi"- Ancona- Sod Clinica Ematologica, Ancona
  - Area Vasta N. 5 Ascoli Piceno - S. Benedetto Del Tronto, Presidio Ospedaliero Av5 Osp. Gen. Prov.Le "C.G.Mazzoni" - Uoc Ematologia, Ascoli Piceno
  - Asl Di Asti, Ospedali Riuniti - Presidio Ospedaliero Cardinal G. Massaia - Sc Oncologia, Asti
  - Asst Degli Spedali Civili Di Brescia - Uo Ematologia, Brescia
  - AO Brotzu, PO A.Businco - SC Ematologia e CTMO, Cagliari
  - Ctc U.O Di Ematologia Con Trapianto Di Midollo Osseo - Catania, Catania
  - Ao Di Catanzaro "Pugliese-Ciaccio", Presidio Ospedaliero "Ciaccio - de Lellis" - Ematologia, Catanzaro
  - Aou Careggi - Firenze - Sod Ematologia, Florence
  - I.R.S.T. Srl Irccs - Meldola - Sc Oncologia Medica, Meldola
  - Ao Ospedali Riuniti "Papardo Piemonte" - Po Papardo - Messina - Sc Ematologia, Messina
  - ASST Grande Ospedale Metropolitano Niguarda - SC Ematologia, Milan
  - Fondazione Irccs "Istituto Nazionale Tumori" - Milano - Sc Ematologia, Milan
  - Fondazione Irccs Ca' Granda, Ospedale Maggiore Policlinico - Milano - Ematologia - Padiglione Marcora, Milan
  - Irccs Ospedale S. Raffaele - Milano - Unità Neoplasie Linfocitarie B, Milan
  - Aou Di Modena - Sc Ematologia, Modena
  - Aou Federico Ii - Napoli - Uoc Ematologia, Napoli
  - Ao Ospedali Riuniti Villa Sofia Cervello - Palermo - Uo Ematologia Con Utmo, Palermo
  - Aou Policlinico P. Giaccone - Palermo - Uo Ematologia, Palermo
  - Aou Di Parma - Sc Ematologia E Centro Trapianti Midollo Osseo, Parma
  - Fondazione Ircss Policlinico San Matteo - Pavia - Uo Ematologia, Pavia
  - Asl Di Piacenza - Ospedale "Guglielmo Da Saliceto" - Ematologia E Centro Trapianti, Piacenza
  - Ao Regionale S. Carlo - Potenza - Sic Ematologia, Potenza
  - Ausl Di Reggio Emilia - Arcispedale Santa Maria Nuova - Irccs - Sc Ematologia, Reggio Emilia
  - Ausl Della Romagna, Ospedale "Infermi" - Rimini - Uo Ematologia, Rimini
  - C.R.O.B. - I.R.C.C.S. - Rionero in Volture - Uoc Ematologia, Rionero in Vulture
  - Aou Policlinico Tor Vergata - Roma - Uoc Trapianto Cellule Staminali, Roma
  - AOU Policlinico Tor Vergata - UOC Trapianto cellule staminali, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli Irccs - Roma - Area Ematologica, Roma
  - Policlinico Universitario Campus Bio Medico - Roma - Uoc Ematologia E Trapianto Di Cellule Staminali, Roma
  - Università Degli Studi Di Roma "Sapienza" - Dipartimento Di Medicina Traslazionale E Di Precisione - U.O.C. Ematologia, Roma
  - A.O.U. Senese - Policlinico "Le Scotte" - UOC EMATOLOGIA E TRAPIANTI, Siena
  - AOU Città della Salute e della Scienza, Ospedale S.Giovanni Battista Molinette - SC Ematologia, Torino
  - Unità Operativa Di Ematologia - Presidio Ospedaliero Di Treviso - Azienda Ulss N.2 Marca Trevigiana, Treviso
  - Asui Di Udine - Presidio Ospedaliero "Santa Maria Della Misericordia" - Clinica Ematologica, Udine
  - Aou Integrata Di Verona, Policlinico G.B. Rossi - Uoc Ematologia, Verona
  - Aulss 8 Berica - Ospedale Di Vicenza - Uoc Ematologia, Vicenza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: GIMEMA Foundation website — http://www.gimema.it